CLINICAL TRIAL: NCT02281123
Title: Study of the Prognostic Value of Musculoskeletal Ultrasound in Adults With Chikungunya
Acronym: EchoCHIK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 14/B/03; 2014-A00875-42 (Other: ANSM)
Record Dates: First submitted 2014-10-29; First posted 2014-11-03 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Infected by Chikungunya Virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient suspected of being infected by chikungunya: Patient (>= 45 ans) suspect d'infection par le virus du chikungunya et présentant des symptomes depuis moins de 10 jours
  Interventions: Other: SF36 (QQoL)

INTERVENTIONS:
Other: SF36 (QQoL) — use of quality of life questionnaire (SF 36) ( at enrollment visit, at 3 month, at 6 month and at12 month for the following visits)

SUMMARY:
Chikungunya is a viral disease transmitted by mosquitoes whose clinical feature is the early joint damage. Approximately 8% of patients have chronic arthropathy resembling to the rheumatoid polyarthritis. The EchoCHIK study we propose is in the context of the epidemic in Martinique which began in January 2014. It should give a better understanding of arthritis and juxtaarticular of CHIK and look for signs that may allow ultrasound predict the evolution of chronic arthropathy of CHIK.

ELIGIBILITY:
Inclusion Criteria:

1. Age at onset of symptoms ≥ 45 years
2. Seen in consultation at the University Hospital of Fort-de-France
3. Suspected chikungunya infection (fever and sudden onset of joint pain affecting the wrists, hands, ankles or knees)
4. Duration of symptoms suggestive of infection chikungunya less than or equal to 10 days
5. Presence of joint pain on the day of inclusion
6. No history of inflammatory arthritis
7. Absence of steroidal or non-steroidal anti-inflammatory drugs taken within two weeks prior to inclusion
8. Ability to participate in the study throughout its duration (12 months)
9. Patient affiliated or beneficiary of a social health care.
10. Acceptance to participate in the study and monitoring proposed and signed informed consent

Exclusion Criteria:

1. Age at onset of symptoms <45 years
2. Duration of symptoms suggestive of chikungunya for more than 10 days
3. Lack of joint pain on the day of inclusion
4. History of inflammatory arthritis Nonsteroidal anti-inflammatory drugs or
5. Taking in the two weeks preceding the inclusion
6. Inability to participate in the study throughout its duration (12 months)
7. Patient is not affiliated or beneficiary of a social health care.
8. Refusal to participate in the study or to sign a consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will be done among the patients from the Fort-de-France hospital and came for a suspected infection by the chikungunya virus
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Presence of sonographic signs observed during the initial scan: periarticular infiltration, effusion, positive Doppler, erosions. | enrollement visit
  Progression to chronic form defined by the persistence or recurrence of muscle symptoms (myalgia) and joints (arthralgia, arthritis) more than two months after the onset of symptoms of acute phase.

SECONDARY OUTCOMES:
Presence of clinical and sonographic signs observed at each visit: arthralgia, arthritis clinics, periarticular infiltration, effusion, positive Doppler erosions. | 1 month, 3 month, 6 month and 12 month after the first symptoms of infection by chikungunya virus

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Brunier-Agot, MD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

REFERENCES:
- [Background] Pialoux G, Gauzere BA, Jaureguiberry S, Strobel M. Chikungunya, an epidemic arbovirosis. Lancet Infect Dis. 2007 May;7(5):319-27. doi: 10.1016/S1473-3099(07)70107-X. PMID 17448935
- [Background] Fourie ED, Morrison JG. Rheumatoid arthritic syndrome after chikungunya fever. S Afr Med J. 1979 Jul 28;56(4):130-2. PMID 494034
- [Background] Kennedy AC, Fleming J, Solomon L. Chikungunya viral arthropathy: a clinical description. J Rheumatol. 1980 Mar-Apr;7(2):231-6. PMID 7373626
- [Background] Brighton SW, Prozesky OW, de la Harpe AL. Chikungunya virus infection. A retrospective study of 107 cases. S Afr Med J. 1983 Feb 26;63(9):313-5. PMID 6298956
- [Background] Simon F, Parola P, Grandadam M, Fourcade S, Oliver M, Brouqui P, Hance P, Kraemer P, Mohamed AA, de Lamballerie X, Charrel R, Tolou H. Chikungunya infection: an emerging rheumatism among travelers returned from Indian Ocean islands. Report of 47 cases. Medicine (Baltimore). 2007 May;86(3):123-137. doi: 10.1097/MD/0b013e31806010a5. PMID 17505252
- [Background] Taubitz W, Cramer JP, Kapaun A, Pfeffer M, Drosten C, Dobler G, Burchard GD, Loscher T. Chikungunya fever in travelers: clinical presentation and course. Clin Infect Dis. 2007 Jul 1;45(1):e1-4. doi: 10.1086/518701. Epub 2007 May 23. PMID 17554689
- [Background] Bouquillard E, Combe B. A report of 21 cases of rheumatoid arthritis following Chikungunya fever. A mean follow-up of two years. Joint Bone Spine. 2009 Dec;76(6):654-7. doi: 10.1016/j.jbspin.2009.08.005. PMID 19945329
- [Background] Larrieu S, Pouderoux N, Pistone T, Filleul L, Receveur MC, Sissoko D, Ezzedine K, Malvy D. Factors associated with persistence of arthralgia among Chikungunya virus-infected travellers: report of 42 French cases. J Clin Virol. 2010 Jan;47(1):85-8. doi: 10.1016/j.jcv.2009.11.014. Epub 2009 Dec 8. PMID 20004145
- [Background] Ribera A, Degasne I, Jaffar Bandjee MC, Gasque P. [Chronic rheumatic manifestations following chikungunya virus infection: clinical description and therapeutic considerations]. Med Trop (Mars). 2012 Mar;72 Spec No:83-5. French. PMID 22693935
- [Background] Manimunda SP, Vijayachari P, Uppoor R, Sugunan AP, Singh SS, Rai SK, Sudeep AB, Muruganandam N, Chaitanya IK, Guruprasad DR. Clinical progression of chikungunya fever during acute and chronic arthritic stages and the changes in joint morphology as revealed by imaging. Trans R Soc Trop Med Hyg. 2010 Jun;104(6):392-9. doi: 10.1016/j.trstmh.2010.01.011. Epub 2010 Feb 19. PMID 20171708
- [Background] Gerardin P, Fianu A, Michault A, Mussard C, Boussaid K, Rollot O, Grivard P, Kassab S, Bouquillard E, Borgherini G, Gauzere BA, Malvy D, Breart G, Favier F. Predictors of Chikungunya rheumatism: a prognostic survey ancillary to the TELECHIK cohort study. Arthritis Res Ther. 2013 Jan 9;15(1):R9. doi: 10.1186/ar4137. PMID 23302155
- See also: A destructive arthropathy following Chikungunya virus arthritis--a possible association — http://www.biomedcentral.com/1471-2334/9/200
- See also: Destructive arthritis in a patient with chikungunya virus infection with persistent specific IgM antibodies — http://www.biomedcentral.com/1471-2334/9/200
- See also: Post-Epidemic Chikungunya Disease on Reunion Island: Course of Rheumatic Manifestations and Associated Factors over a 15-Month Period — http://www.plosntds.org/article/info%3Adoi%2F10.1371%2Fjournal.pntd.0000389